CLINICAL TRIAL: NCT05964348
Title: REGISTRY for the Use of a Software for Automatic Detection of the Evolution of Aneurysmal Volume and Graft Migration After EVAR (EndoVascular Aneurysm Repair)
Acronym: AI-EVAR-FOLLOW
Status: Withdrawn | Type: Observational
Why Stopped: the study was no longer of scientific interest, and other publications rendered it obsolete
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Nurea (Industry)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2022/66
Record Dates: First submitted 2023-05-11; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Aneurysm Aortic
Keywords: Abdominal Aortic Aneurysm; CT scan; Semi-automated analyses; Software
MeSH Terms: conditions — Aortic Aneurysm; Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with infrarenal abdominal aortic aneurysms: Patient with infrarenal abdominal aortic aneurysms treated with EVAR
  Interventions: Procedure: CT-Scan

INTERVENTIONS:
Procedure: CT-Scan — semi-automated analyse by anatomical landmarks with a dedicated fully automated software

SUMMARY:
The objective of this registry is to find and validate a correlation between morphological indicators such as volume sac evolution, graft migration or length between anatomical landmarks with aneurysm rupture risk or complications such as endoleaks requiring re-intervention… Secondary objectives are the validation of the reproducibility and accuracy of a dedicated fully automated software enabling Abdominal Aortic Aneurysm (AAA) segmentation to measure AAA diameter, volume evolution and growth over time, proximal and distal sealing zones analyze as well as device migration and integrity after EVAR on computed tomography angiography (CTA). This validation is in comparison with semi-automated analyse controlled by physician.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age
* Infra-renal Abdominal Aortic Aneurysm (AAA) treated with EVAR

  * ≥50mm
  * or ≥5mm increase in 6 months
  * or surviving Ruptured AAA
* legal capacity to make own decisions, informed of the nature of the registry, has signed non opposition form available for set-up and proper implementation of follow-up visits throughout the duration of the registry

Exclusion Criteria:

* Advancing Alzheimer's disease or socially dependent patient
* Opposition to the use of their data for this research
* Life expectancy supposed to be inferior to 2 years Pregnant female

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male or female ≥18 years of age with an Infra-renal Abdominal Aortic Aneurysm treated with endovascular treatment, ≥50mm, or ≥5mm increase in 6 months or surviving Ruptured AAA
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Collection of the different events and complications of the aneurysm post EVAR | Month 1
  Collection of the different events and complication occurred after the EVAR (post-operative (up to one month), 3, 6 and 12 months). The collection will be use to correlate with the measurement of the morphological indicators collected at the different time frame of the study
Collection of the different events and complications of the aneurysm post EVAR | Month 3
  Collection of the different events and complication occurred after the EVAR (post-operative (up to one month), 3, 6 and 12 months). The collection will be use to correlate with the measurement of the morphological indicators collected at the different time frame of the study
Collection of the different events and complications of the aneurysm post EVAR | Month 6
  Collection of the different events and complication occurred after the EVAR (post-operative (up to one month), 3, 6 and 12 months). The collection will be use to correlate with the measurement of the morphological indicators collected at the different time frame of the study
Collection of the different events and complications of the aneurysm post EVAR | Month 12
  Collection of the different events and complication occurred after the EVAR (post-operative (up to one month), 3, 6 and 12 months). The collection will be use to correlate with the measurement of the morphological indicators collected at the different time frame of the study
Measurement of aneurysm sac volume evolution | Month 1
  Measurement of the aneurysm sac volume in cc on the CT scans available
Measurement of aneurysm sac volume evolution | Month 3
  Measurement of the aneurysm sac volume in cc on the CT scans available
Measurement of aneurysm sac volume evolution | Month 6
  Measurement of the aneurysm sac volume in cc on the CT scans available
Measurement of aneurysm sac volume evolution | Month 12
  Measurement of the aneurysm sac volume in cc on the CT scans available
Measurement of morphological neck characteristics | Month 6 before intervention
  Measurement of the morphological neck characteristics in mm on the CT scans available
Measurement of morphological neck characteristics | Month 1
  Measurement of the morphological neck characteristics in mm on the CT scans available
Measurement of morphological neck characteristics | Month 3
  Measurement of the morphological neck characteristics in mm on the CT scans available
Measurement of morphological neck characteristics | Month 6
  Measurement of the morphological neck characteristics in mm on the CT scans available
Measurement of morphological neck characteristics | Month 12
  Measurement of the morphological neck characteristics in mm on the CT scans available
Measurement of graft migration | 6 months before intervention
  Measurement of the graft migration if existing on the CT scans available
Measurement of graft migration | Month 1
  Measurement of the graft migration if existing on the CT scans available
Measurement of graft migration | Month 3
  Measurement of the graft migration if existing on the CT scans available
Measurement of graft migration | Month 6
  Measurement of the graft migration if existing on the CT scans available
Measurement of graft migration | Month 12
  Measurement of the graft migration if existing on the CT scans available
Measurement of length between anatomical points evolution | 6 months before intervention
  Measurement of the length between anatomical points evolution of the aneurysm in mm on the CT scans available.
Measurement of length between anatomical points evolution | Month 1
  Measurement of the length between anatomical points evolution of the aneurysm in mm on the CT scans available.
Measurement of length between anatomical points evolution | Month 3
  Measurement of the length between anatomical points evolution of the aneurysm in mm on the CT scans available.
Measurement of length between anatomical points evolution | Month 6
  Measurement of the length between anatomical points evolution of the aneurysm in mm on the CT scans available.
Measurement of length between anatomical points evolution | Month 12
  Measurement of the length between anatomical points evolution of the aneurysm in mm on the CT scans available.

SECONDARY OUTCOMES:
Repeatability between one senior and one junior surgeon (inter observer variability) for the Semi-automatic segmentation | Month
  Descriptive analysis of the semi-automatic segmentation for the junior and senior surgeon by overlaps metric analysis
Repeatability between one senior and one junior surgeon (inter observer variability) for the Semi-automatic segmentation | 6 months before intervention
  Descriptive analysis of the semi-automatic segmentation for the junior and senior surgeon by overlaps metric analysis
Repeatability between one senior and one junior surgeon (inter observer variability) for the Semi-automatic segmentation | Month 1
  Descriptive analysis of the semi-automatic segmentation for the junior and senior surgeon by overlaps metric analysis
Repeatability between one senior and one junior surgeon (inter observer variability) for the Semi-automatic segmentation | Month 3
  Descriptive analysis of the semi-automatic segmentation for the junior and senior surgeon by overlaps metric analysis
Repeatability between one senior and one junior surgeon (inter observer variability) for the Semi-automatic segmentation | Month 6
  Descriptive analysis of the semi-automatic segmentation for the junior and senior surgeon by overlaps metric analysis
Repeatability between one senior and one junior surgeon (inter observer variability) for the Semi-automatic segmentation | Month 12
  Descriptive analysis of the semi-automatic segmentation for the junior and senior surgeon by overlaps metric analysis
Repeatability between measures (intra observer variability) | 6 months before intervention
  Descriptive analysis of the different measurements by overlaps metric analysis
Repeatability between measures (intra observer variability) | Month 1
  Descriptive analysis of the different measurements by overlaps metric analysis
Repeatability between measures (intra observer variability) | Month 3
  Descriptive analysis of the different measurements by overlaps metric analysis
Repeatability between measures (intra observer variability) | Month 6
  Descriptive analysis of the different measurements by overlaps metric analysis
Repeatability between measures (intra observer variability) | Month 12
  Descriptive analysis of the different measurements by overlaps metric analysis
Average time for segmentation (sec) | 6 months before intervention
  The time for segmentation by junior/senior surgeon and software is recorded
Average time for segmentation (sec) | Month 1
  The time for segmentation by junior/senior surgeon and software is recorded
Average time for segmentation (sec) | Month 3
  The time for segmentation by junior/senior surgeon and software is recorded
Average time for segmentation (sec) | Month 6
  The time for segmentation by junior/senior surgeon and software is recorded
Average time for segmentation (sec) | Month 12
  The time for segmentation by junior/senior surgeon and software is recorded
Average time for segmentation in comparison with semi-automated segmentation | 6 months before intervention
  Description of the average time between the different techniques.
Average time for segmentation in comparison with semi-automated segmentation | Month 1
  Description of the average time between the different techniques.
Average time for segmentation in comparison with semi-automated segmentation | Month 3
  Description of the average time between the different techniques.
Average time for segmentation in comparison with semi-automated segmentation | Month 6
  Description of the average time between the different techniques.
Average time for segmentation in comparison with semi-automated segmentation | Month 12
  Description of the average time between the different techniques.
Total Volume measurement of AAA | 6 months before intervention
  Description of the volume measurement of the AAA with the following items:
  * Volume circulating
  * Intraluminal thrombus volume
  * Calcification volume
Total Volume measurement of AAA | Month 1
  Description of the volume measurement of the AAA with the following items:
  * Volume circulating
  * Intraluminal thrombus volume
  * Calcification volume
Total Volume measurement of AAA | Month 3
  Description of the volume measurement of the AAA with the following items:
  * Volume circulating
  * Intraluminal thrombus volume
  * Calcification volume
Total Volume measurement of AAA | Month 6
  Description of the volume measurement of the AAA with the following items:
  * Volume circulating
  * Intraluminal thrombus volume
  * Calcification volume
Total Volume measurement of AAA | Month 12
  Description of the volume measurement of the AAA with the following items:
  * Volume circulating
  * Intraluminal thrombus volume
  * Calcification volume

CONTACTS AND LOCATIONS:
Overall Officials: Eric Ducasse, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Service de Chirurgie Vasculaire, Hôpital Pellegrin-tripode, CHU de Bordeaux, Bordeaux, France